CLINICAL TRIAL: NCT04016376
Title: Cluster-Randomized, Prospective Assessment of Postoperative Pain Management in Patients Undergoing Bilateral Mastectomy With Immediate Reconstruction With Tissue Expander (BMWRw/TE) Using Preoperative Paravertebral (PVB), Serratus+PECS-1, or PVB+PECS-1 Nerve Blocks
Brief Title: Study of Nerve Block Pain Management in Patients Undergoing a Double Mastectomy With Immediate Reconstruction
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-238
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Breast Cancer Female
Keywords: Mastectomy; Double Mastectomy; Mastectomy with reconstruction; Double mastectomy with reconstruction; Double mastectomy with immediate reconstruction; Mastectomy with immediate reconstruction; Memorial Sloan Kettering Cancer Center; 19-238
MeSH Terms: conditions — Breast Neoplasms | interventions — PVB protocol

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to 1 of 3 groups (approximately n=500 patients per group) of standard of care preoperative nerve blocks consisting of either: i) PVB, ii) serratus+PECS-1, or iii) PVB+PECS-1. Each group will receive ropivacaine or bupivacaine +/- clonidine (0.5 - 1 mcg/kg not to exceed a total of 100 mcg) +/- dexamethasone (up to 4 mg) in one of three routine nerve block approaches prior to surgical procedure as is current standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PVB (Experimental): Patient will be placed in the prone, lateral, or sitting position. With an ultrasound probe placed in the parasagittal or transverse position, the paravertebral space will be identified. Injections will be done in an in-plane manner relative to the ultrasound probe. Local anesthesia will be injected to cover T1-T6 dermatomes.
  Interventions: Drug: PVB Protocol
- PVB + PECS-1 (Experimental): Patient will be placed in the prone, lateral, or sitting position. With an ultrasound probe placed in the parasagittal or transverse position, the paravertebral space will be identified. Injections will be done in an in-plane manner relative to the ultrasound probe. Local anesthesia will be injected to cover T1-T6 dermatomes.
  For PECS-1, the patient will be placed in the supine position with an ultrasound probe placed inferolaterally starting at the mid-clavicular level the pectoralis major and minor will be identified. Injection of local anesthesia will be performed between the pectoralis major and minor.
  Interventions: Drug: PVB Protocol; Drug: PECS-1
- Serratus + PECS-1 (Experimental): For PECS-1, the patient will be placed in the supine position with an ultrasound probe placed inferolaterally starting at the mid-clavicular level the pectoralis major and minor will be identified. Injection of local anesthesia will be performed between the pectoralis major and minor.
  For the serratus block, the patient will be placed in the supine or lateral decubitus position and with an ultrasound probe, in the parasagittal plane, the serratus muscles will be identified. Injections will be done in-plane below the serratus anterior.
  Interventions: Drug: PECS-1; Drug: Serratus

INTERVENTIONS:
Drug: PVB Protocol — Patient will be placed in the prone, lateral, or sitting position. With an ultrasound probe placed in the parasagittal or transverse position, the paravertebral space will be identified. Injections will be done in an in-plane manner relative to the ultrasound probe. Local anesthesia will be injected to cover T1-T6 dermatomes.
  Arms: PVB; PVB + PECS-1
Drug: PECS-1 — For PECS-1, the patient will be placed in the supine position with an ultrasound probe placed inferolaterally starting at the mid-clavicular level the pectoralis major and minor will be identified. Injection of local anesthesia will be performed between the pectoralis major and minor
  Arms: PVB + PECS-1; Serratus + PECS-1
Drug: Serratus — For the serratus block, the patient will be placed in the supine or lateral decubitus position and with an ultrasound probe, in the parasagittal plane, the serratus muscles will be identified. Injections will be done in-plane below the serratus anterior.
  Arms: Serratus + PECS-1

SUMMARY:
The purpose of this study is to determine if the injection site or sites used for administering pain medication (nerve blocks) before a double mastectomy with immediate reconstruction with tissue expanders reduce the need for pain medication after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients >/= 18 years old
* Undergoing Bilateral Mastectomy with immediate reconstruction (BMw/IR)
* Scheduled for surgery at Josie Robertson Surgical Center (JRSC)
* Must be appropriate for an agree to receive a nerve block
* Must be appropriate for randomization
* Able to read and speak English
* Willing and able to provide written informed consent

Exclusion Criteria:

* None applicable, as exclusion occurs prior to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1507 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Compare preoperative nerve blocks between a combination of nerve blocks and PVB alone to decrease postoperative opioid consumption | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Hanae Tokita, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Tokita HK, Assel MJ, Serafin J, Lin E, Sarraf L, Masson G, Nelson JA, Moo TA, McCready T, Vakassi C, Hingula L, Jackson J, Horine S, Baqai-Stern A, Lewis A, Nadav D, Teng H, Kim J, Hagen J, Scanlon M, Puttanniah V, Legler A, Gauran C, Simon BA, Vickers A. Paravertebral or Serratus Anterior Plane Block Combined with Interpectoral Blocks versus Paravertebral Block for Mastectomy: A Cluster-randomized Trial of 1,507 Patients. Anesthesiology. 2026 Feb 1;144(2):379-389. doi: 10.1097/ALN.0000000000005842. Epub 2025 Nov 10. PMID 41212546
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org